CLINICAL TRIAL: NCT04056962
Title: Tacrolimus for the Treatment of Superficial Kaposiform Hemangioendothelioma and Tufted Angioma：a Randomized Controlled Study
Brief Title: Tacrolimus for the Treatment of Superficial Kaposiform Hemangioendothelioma and Tufted Angioma
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: West China Hospital (Other)
Responsible Party: Principal Investigator, Yi Ji, Doctor of Philosophy, Doctor of Medicine, West China Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 813
Record Dates: First submitted 2019-08-11; First posted 2019-08-14 (Actual); Last update posted 2024-05-07 (Actual); Status verified 2024-05

CONDITIONS: Tacrolimus, Kaposiform Hemangioendothelioma, Tufted Angioma
MeSH Terms: conditions — Kaposiform Hemangioendothelioma; Tufted angioma

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- patients treated with tacrolimus 0.03% ointment (Experimental): patients treated with tacrolimus 0.03% ointment
  Interventions: Drug: Tacrolimus ointment
- patients treated with tacrolimus 0.1% ointment (Active Comparator): patients treated with tacrolimus 0.1% ointment
  Interventions: Drug: Tacrolimus ointment

INTERVENTIONS:
Drug: Tacrolimus ointment — topical application of tacrolimus at different concentrations for treatment of superficial Kaposiform hemangioendothelioma (KHE) and tufted angioma (TA).

SUMMARY:
The aim of this study was to evaluate the efficacy and safety of topical application of tacrolimus at different concentrations for superficial Kaposiform hemangioendothelioma (KHE) and tufted angioma (TA).

DETAILED DESCRIPTION:
Kaposiform hemangioendothelioma (KHE) and tufted angiomas (TA) are rare vascular tumors, which are apparent predominantly in infancy or early childhood. Currently, no standard treatment regimens exist for KHE/TA. The aim of this study was to evaluate the efficacy and safety of topical application of tacrolimus at different concentrations for superficial Kaposiform hemangioendothelioma (KHE) and tufted angioma (TA).

ELIGIBILITY:
Inclusion Criteria:

* Children with superficial Kaposiform hemangioendothelioma (KHE) and tufted angioma (TA)

Exclusion Criteria:

* Hypersensitivity to Tacrolimus Mucosal Kaposiform hemangioendothelioma (KHE) and tufted angioma (TA)

Ages: 0 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 50 (Estimated)
Dates: Start 2019-09-01 (Actual); Primary Completion 2024-08-30 (Estimated); Study Completion 2024-10-28 (Estimated)

PRIMARY OUTCOMES:
reduction in the size of the lesion | 2.5 years
  Therapeutic effect is evaluated by reduction in the size of the tumor measured by centimeters.

SECONDARY OUTCOMES:
Rate of Adverse events | 2.5 years
  using the measurement of ratio to evaluate the rate of adverse events of topical application of tacrolimus (such as ratio of Acne vulgaris, pruritis and rash etc.).

CONTACTS AND LOCATIONS:
Overall Officials: Yi Ji, Principal Investigator — West China Hospital
Locations (1):
- West China Hospital of Sichuan University, Chengdu, Sichuan, China

IPD SHARING:
Plan to Share IPD: No